CLINICAL TRIAL: NCT06536166
Title: Blocking Interferon-γ by Ruxolitinib for Treating Inclusion Body Myositis: a Phase IIb Trial
Brief Title: Ruxolitinib Treatment in Inclusion Body Myositis
Acronym: BIGTIM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP220829
Record Dates: First submitted 2024-07-26; First posted 2024-08-02 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Inclusion Body Myositis, Sporadic
Keywords: Inclusion body myositis; Idiopathic immune myopathy; JAK-inhibitor; Ruxolitinib
MeSH Terms: conditions — Myositis, Inclusion Body | interventions — ruxolitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Randomization in experimental group.
  Interventions: Drug: Ruxolitinib
- Control group (Placebo Comparator): Randomization in control group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ruxolitinib — IBM patients treated by ruxolitinib (JAKAVI®), 15mg per os, twice a day, during 12 months.
  Arms: Experimental group
Drug: Placebo — IBM patients treated by placebo, twice a day, during 12 months.
  Arms: Control group

SUMMARY:
Refer to the "Detailed Description" section.

DETAILED DESCRIPTION:
A Phase II/III Randomized, Double-blind, Placebo-controlled, Multicenter Study to Determine the Efficacy and Safety of Ruxolitinib in the Treatment of Subjects with Inclusion Body Myositis (IBM) IBM is the most frequent idiopathic immune myopathy (IIM) over age 45, pathologically characterized by the combination of intramuscular inflammation and degenerative features. It differs from other IIMs by its chronic evolution and refractoriness to common immunomodulatory drugs leading to marked disability and poor quality of life. Histological and molecular analyses of muscle biopsies from IBM patients showed intense muscular type II interferon (IFNγ) signature, stronger than observed in other IIMs. In vitro and in vivo experimental studies showed that IFNγ exerts myosuppressive effects through JAK/STAT pathway activation mimicking the degenerative features observed in IBM, and that these effects can be prevented by JAK-inhibitor ruxolitinib.

Hypothesis/Objective : Ruxolitinib could be an effective therapy for IBM. Objective is to evaluate its therapeutic effects in IBM.

Method : Comparative, multicenter, randomized, parallel-group, superiority, placebo-controlled, double-blind, phase 2 trial. 60 IBM patients able to walk during at least 6mn will be randomized in two groups (30/group) and received either ruxolitinib 15mgx2/d or placebo during 1 yr. Evaluation includes 6MWT, muscle strength quantification, functional scales, respiratory functional test and muscle MRI.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 45 years
* Effective contraception for the duration of the clinical trial for fertile women of childbearing age
* Defined diagnosis of IBM according to data-derived criteria (Llyod et al, 2014): Patient must fulfill the three following criteria for being diagnosed as IBM: (1) finger flexor or quadriceps weakness; and (2) muscle biopsy showing endomysial inflammation; and (3) muscle biopsy showing invasion of nonnecrotic muscle fibers or rimmed vacuoles
* To be able to walk 6 min without assistance from another person (external assist devices permitted [e.g., canes, walkers, or rollators])
* Patient informed and having signed the consent for participation, possibly assisted by a trusted person

Exclusion Criteria:

* Pregnancy or breastfeeding
* Patient under guardianship, curatorship, safeguard of justice or deprived of liberty
* Patient with cognitive disorders or unable, according to the investigator, to understand the study and/or to give informed consent
* Quadriceps weakness (manual muscle testing, MRC) below or equal 1
* Forced vital capacity (FVC) or forced expiratory volume (FEV) < 50% of predicted value
* Concomitant use of immunomodulatory drugs including previous treatment with JAK inhibitor, or medications acting on muscle anabolism or catabolism
* Live vaccine within the 4 weeks before starting treatment
* Comorbidity or active chronic disease which contraindicate ruxolitinib:

  * Lipid parameters abnormalities/elevations
  * Severe renal impairment (stage 4) and end-stage renal disease (stage 5)
  * Hepatic impairment
  * Cytopenia
  * Recent history (<6 months) of cardiovascular or thromboembolic disease (documented coronaropathy or hospitalization for acute arterial thrombosis or stroke or deep venous thrombosis or pulmonary embolism)
  * Active smoking more than 20 pack-years or history of respiratory or skin cancer or recent history (<6 months) of other neoplastic disease
  * Very high cardiovascular risk (red color) at SCORE 2 in case of recent history (<6 months) of cardiovascular or thromboembolic disease and non-controlled cardiovascular risk factors
  * History of Stevens-Johnson's syndrome or Lyell's syndrome
* Active SARS-CoV-2 infection (patient can be included once infection resolved)
* Any medical condition which limits the ability of participant to participate in study
* Necessity to use a drug incompatible with ruxolitinib
* Hypersensitivity to the IMP's active substance (ruxolitinib) or to any of the excipients
* Non-affiliation to a social security scheme or to another social protection scheme, patient on state medical aid
* Foreseeable inability, according to the investigator, to participate in all the visits, treatments and measures provided for in the protocol
* Concomitant participation in another clinical trial on medical product for human use, to a clinical investigation on a medical device, to interventional study involving human participants or in the exclusion period at the end of a previous clinical trial on medical product for human use, a clinical investigation on a medical device, or study involving human participants.

Participation in non-interventional research is permitted.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2028-06-10 (Estimated); Study Completion 2028-09-10 (Estimated)

PRIMARY OUTCOMES:
6 minutes-walk distance (6MWT): A distance walked in 6 min. superior in treated patients compared to placebo group | 12 months
  The 6MWT is performed in a corridor, between two cones separated by a distance of 25 m.

SECONDARY OUTCOMES:
Adverse events (safety and tolerability) of ruxolitinib in IBM patients | Through study completion that is to say 15 months
  Adverse events collected according to the MedDRA classification
Therapeutic muscular efficacy of ruxolitinib on muscle strength | Until last consultation that is to say 12 months
  Quantification of muscle strength using dynamometer
Therapeutic muscular efficacy of ruxolitinib on overall muscle status | Until last consultation that is to say 12 months
  Measurement of overall muscle status using scales and serum creatine kinase (CK) levels
Respiratory ability | 12 months
  Forced vital capacity (FVC) measurement
Evaluate swallowing using Swallowing Disturbance Questionnaire (SDQ) | 12 months
  Measurement of the swallowing disorders via Swallowing Disturbance Questionnaire (SDQ). 15 items. Overall score from 0,5 to 44,5. The score increase with the swallowing disorders.
Lower limb quantification of fat replacement of muscle tissue, residual muscle tissue and markers of disease activity using MRI | 12 months
  Measurement of the differences in fat fraction value calculated on thigh Dixon MRI pictures
Evaluate quality of life using Health Assessment Questionnaire without Disability Index (HAQ-DI) | 12 months
  Measurement of the difference in the quality of life measured by Health Assessment Questionnaire without Disability Index (HAQ-DI). 8 dimensions rated from 0 (without any difficulty) to 3 (unable to do). Overall score from 0 to 3. The higher the score, the lower the quality of life.
Evaluate quality of life using Duke health profile | 12 months
  Measurement of the difference in the quality of life measured by Duke health profile - The Duke. 10 dimensions. Overall score from 0 to 100. The score increase with the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: François Jérôme AUTHIER, Pr, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (16):
- France (16):
  - Hôpital Pellegrin - Tripode, CHU de Bordeaux, Bordeaux, France
  - Hôpital Pierre Wertheimer, CHU de Lyon, Bron, France
  - CHU Caen Normandie, Caen, France
  - Hôpital Henri-Mondor, APHP, Créteil, France
  - Hôpital Raymond Poincaré, APHP, Garches, France
  - Hôpital Roger Salengro, CHU de Lille, Lille, France
  - Hôpital Dupuytren, CHU de Limoges, Limoges, France
  - Hôpital de la Timone, APHM, Marseille, France
  - CHU Nancy, Nancy, France
  - Hôtel-Dieu, CHU Nantes, Nantes, France
  - Hôpital Pasteur, CHU de Nice, Nice, France
  - Hôpital Pitié-Salpêtrière, APHP, Paris, France
  - Hôpital Christian Cabrol, CHU Reims, Reims, France
  - Hôpital Bellevue, CHU Saint-Etienne, Saint-Etienne, France
  - Hôpital de Hautepierre, Hôpitaux Universitaires de Strasbourg, Strasbourg, France
  - Hôpital Pierre-Paul Riquet, CHU de Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No
Datas are own by assistance publique - hopitaux de paris, please contact sponsor for further information.